CLINICAL TRIAL: NCT02062671
Title: Renal Sympathetic Denervation for Reduction of Pain and Improvement of Insulin Sensitivity in Adult Polycystic Kidney Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Odense University Hospital (Other)
Responsible Party: Principal Investigator, Hans Dieperink, Head of Department, MD, Odense University Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: RePKID; S-20130085 (Registry Identifier: De Videnskabsetiske komitéer for Region Syddanmark)
Record Dates: First submitted 2014-02-12; First posted 2014-02-14 (Estimated); Last update posted 2014-02-14 (Estimated); Status verified 2014-02

CONDITIONS: Adult Polycystic Kidney Disease
Keywords: ADPKD; denervation; renal denervation
MeSH Terms: conditions — Polycystic Kidney, Autosomal Dominant

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- immediate renal denervation (Experimental): immediate renal denervation
  Interventions: Procedure: renal denervation
- delayed renal denervation (Active Comparator): delayed renal denervation
  Interventions: Procedure: renal denervation

INTERVENTIONS:
Procedure: renal denervation

SUMMARY:
In patients with polycystic kidney disease, pain may be resistant to drug therapy and may reduce quality of life. This study investigate the effect of renal denervation on this pain.

ELIGIBILITY:
Inclusion Criteria:

* Pain limiting daily activities in spite of pain killers, ADPKD

Exclusion Criteria:

* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2014-02; Primary Completion 2015-02 (Estimated); Study Completion 2015-02 (Estimated)

PRIMARY OUTCOMES:
Pain | 6 months
  Pain from VAS

SECONDARY OUTCOMES:
Quality of Life (QoL) | 6 months
  SF-12v2

OTHER OUTCOMES:
kidney function | 6 months
  creatinine clearance

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Nephrology, Odense, Denmark